CLINICAL TRIAL: NCT00498628
Title: A Phase 2, Double-Blind, Placebo Controlled Trial to Assess the Efficacy of Quetiapine Fumarate Extended Release for the Treatment of Alcohol Dependence in Very Heavy Drinkers.
Brief Title: Study of the Effectiveness of Quetiapine for the Treatment of Alcohol Dependency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); AstraZeneca (Industry); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIAAA_DTRR-2007-LITTEN-01
Record Dates: First submitted 2007-07-06; First posted 2007-07-10 (Estimated); Results first posted 2012-05-30 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-02

CONDITIONS: Alcoholism; Alcohol Abuse
Keywords: Alcoholism; Alcohol dependence; Quetiapine
MeSH Terms: conditions — Alcoholism | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Quetiapine fumarate plus medical management
  Interventions: Drug: Quetiapine fumarate
- 2 (Placebo Comparator): Medical management plus placebo comparator
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Quetiapine fumarate — Quetiapine fumarate- taken daily, for 12 weeks
  Other Names: SEROQUEL XR
  Arms: 1
Other: Placebo — Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether quetiapine fumarate extended release is effective in the treatment of alcohol dependence in very heavy drinkers.

DETAILED DESCRIPTION:
This study will investigate quetiapine fumarate XR (SEROQUEL XR®), a dibenzothiazepine derivative, as a potential medication for treating alcohol dependence. The immediate release form of quetiapine fumarate, SEROQUEL XR®, is approved by the FDA for treatment of schizophrenia and acute manic episodes associated with bipolar disorder. The extended release formulation (SEROQUEL XR®) is also approved by the FDA and is undergoing clinical investigation for the treatment of major depressive disorders, schizophrenia, generalized anxiety disorder, and alcohol dependence.

Treatment with other atypical antipsychotics such as clozapine and olanzapine has resulted in decreases in alcohol use in alcohol dependent patients with and without comorbid psychiatric diagnoses. Quetiapine, like clozapine, appears to have efficacy in reducing drug and alcohol use among alcoholics and drug dependent patients with co-morbid psychiatric illness.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65 years old
* DSM-IV diagnosis of current alcohol dependence as supported by SCID Module E
* Report "very heavy" drinking (10 or more drinks per drinking day for men or 8 or more drinks per drinking day for women) at least 40% of the days during the interval from day 31 to 90 prior to the initial screening visit (i.e. a total of 24 days of this 60-day period), with at least one day of "very heavy" drinking occurring within the last 2 weeks before screening
* Seeking treatment for alcohol dependence and desire reduction or cessation of drinking
* Able to verbalize understanding of the consent form, able to provide written informed consent, and verbalize willingness to complete study procedures
* Females of child bearing potential must agree to use of at least one approved method of birth control, or must be surgically sterile or postmenopausal
* Able to take oral medication, willing to adhere to the medication regimen, and willing to return for regular visits
* Able to understand written and oral instructions in English and to complete the questionnaires required by the protocol
* Can complete all psychological assessments required at screening and baseline
* Able to provide evidence of stable residence in the last 2 months prior to randomization, have reasonable transportation arrangements to study site, and have no plans to move within the next 3 months or unresolved legal problems; must provide contact information of family member, spouse, or significant other who can contact subject in case of missed appointment
* Breath alcohol concentration (BAC) equal to 0.00 when s/he signed the informed consent document
* Must have an absolute neutrophil count of 1.5 x 109/L or greater.

Exclusion Criteria:

Please contact site for additional information.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2007-12; Primary Completion 2009-08 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raye Z. Litten, PhD, Study Director — National Institute on Alcohol Abuse and Alcoholism (NIAAA); Margaret E. Mattson, PhD, Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA); Joanne Fertig, PhD, Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (7):
- United States (7):
  - Boston University School of Medicine, Psychiatry Clinical Studies Unit, Boston, Massachusetts
  - Dartmouth Medical School, Dept. of Psychiatry, Lebanon, New Hampshire
  - University of Pennsylvania, Treatment Research Center, Philadelphia, Pennsylvania
  - Brown University Center for Alcohol and Addiction Studies, Providence, Rhode Island
  - White River Junction VA Medical Center, White River Junction, Vermont
  - University of Virginia, Dept. of Psychiatric Medicine, Charlottesville, Virginia
  - University of Virginia, Richmond, Virginia

REFERENCES:
- [Result] Litten RZ, Fertig JB, Falk DE, Ryan ML, Mattson ME, Collins JF, Murtaugh C, Ciraulo D, Green AI, Johnson B, Pettinati H, Swift R, Afshar M, Brunette MF, Tiouririne NA, Kampman K, Stout R; NCIG 001 Study Group. A double-blind, placebo-controlled trial to assess the efficacy of quetiapine fumarate XR in very heavy-drinking alcohol-dependent patients. Alcohol Clin Exp Res. 2012 Mar;36(3):406-16. doi: 10.1111/j.1530-0277.2011.01649.x. Epub 2011 Sep 26. PMID 21950727
- [Derived] Vatsalya V, Kong M, Marsano LM, Kurlawala Z, Chandras KV, Schwandt ML, Ramchandani VA, McClain CJ. Interaction of Heavy Drinking Patterns and Depression Severity Predicts Efficacy of Quetiapine Fumarate XR in Lowering Alcohol Intake in Alcohol Use Disorder Patients. Subst Abuse. 2020 Sep 9;14:1178221820955185. doi: 10.1177/1178221820955185. eCollection 2020. PMID 32963470

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Interested candidates responded by telephone to advertisements at 5 academic centers in the United States between December 2007 and May 2009.
Pre-assignment Details: 218 comprises the Modified Intent To Treat group (MITT)
Groups:
- Quetiapine Fumerate Plus Medical Management: Quetiapine fumarate - target dose 400mg/day plus medical management
- Sugar Pill Plus Medical Management: Medical management plus placebo comparator
Period: Overall Study
Arm/Group | Quetiapine Fumerate Plus Medical Management | Sugar Pill Plus Medical Management
Started | 105 | 113
Completed | 90 | 92
Not Completed | 15 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine Fumerate Plus Medical Management | Sugar Pill Plus Medical Management | Total
Number analyzed (Participants) | 105 | 113 | 218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 105 | 113 | 218
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (9.3) | 45.5 (9.8) | 45.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 26 | 43
  Male | 88 | 87 | 175
Region of Enrollment [Number; unit: participants]
  United States | 105 | 113 | 218

OUTCOME MEASURES:

1. Primary Outcome: Percent Heavy Drinking Days
Description: A heavy drinking day is defined as 5 or more drinks for men and 4 or more drinks for women during a 24 hour period.
Time Frame: Weeks 3 - 11
Population: Intention to Treat
Measure: Least Squares Mean (Standard Error); unit: percentage of heavy drinking days
Arm/Group | Quetiapine Fumerate Plus Medical Management | Sugar Pill Plus Medical Management
Number analyzed (Participants) | 105 | 113
percentage of heavy drinking days | 37.1 (3.5) | 37.9 (3.34)

2. Secondary Outcome: Percent Days Abstinent
Description: Timeline Follow-back drinking data is used to calculate the % of days abstinent per week during Weeks 3-11
Time Frame: Weeks 3-11
Measure: Least Squares Mean (Standard Error); unit: percentage of days abstinent
Arm/Group | Quetiapine Fumerate Plus Medical Management | Sugar Pill Plus Medical Management
Number analyzed (Participants) | 105 | 113
percentage of days abstinent | 49.5 (3.71) | 47.1 (3.54)

3. Secondary Outcome: Drinks Per Drinking Day
Description: Timeline Follow Back daily drinking data used to calculate the weekly mean drinks per drinking day
Time Frame: Study Weeks 3-11
Measure: Least Squares Mean (Standard Error); unit: drinks per drinking day
Arm/Group | Quetiapine Fumerate Plus Medical Management | Sugar Pill Plus Medical Management
Number analyzed (Participants) | 105 | 113
drinks per drinking day | 6.2 (.47) | 6.3 (.45)

4. Secondary Outcome: Drinks Per Day
Description: Timeline Follow Back daily drinking data used to calculate the weekly mean drinks per day
Time Frame: Study Weeks 3-11
Measure: Least Squares Mean (Standard Error); unit: drinks per day
Arm/Group | Quetiapine Fumerate Plus Medical Management | Sugar Pill Plus Medical Management
Number analyzed (Participants) | 105 | 113
drinks per day | 4.3 (0.43) | 4.4 (0.41)

5. Secondary Outcome: Percent Very Heavy Drinking Day
Description: Timeline Follow Back data used to calculate the % of very heavy drinking days per week. Heavy drinking is 10+ drinks per day for females and 12+ drinks per day for males
Time Frame: Study Weeks 3-11
Measure: Least Squares Mean (Standard Error); unit: percentage heavy drinking days
Arm/Group | Quetiapine Fumerate Plus Medical Management | Sugar Pill Plus Medical Management
Number analyzed (Participants) | 105 | 113
percentage heavy drinking days | 16.5 (2.56) | 18.8 (2.44)

6. Secondary Outcome: Percent Subjects Abstinent
Description: Timeline Follow Back data used to calculate the % of subjects that maintained abstinence weeks 3-11.
Time Frame: Study Weeks 3-11
Measure: Count of Participants; unit: Participants
Arm/Group | Quetiapine Fumerate Plus Medical Management | Sugar Pill Plus Medical Management
Number analyzed (Participants) | 105 | 113
Participants | 12 | 12

7. Secondary Outcome: Percent Subjects With no Heavy Drinking Day
Description: Timeline Follow Back data used to calculate the % of subjects that didn't have a heavy drinking day during study weeks 3-11.
Time Frame: Study Weeks 3-11
Measure: Count of Participants; unit: Participants
Arm/Group | Quetiapine Fumerate Plus Medical Management | Sugar Pill Plus Medical Management
Number analyzed (Participants) | 105 | 113
Participants | 17 | 24

8. Secondary Outcome: Drinking Consequences Score
Description: Drinkers Inventory of Consequences (DrInC) - Alcohol-related problems are determined using the DrInC (Miller et al., 1995). The DrInC is a self-administered 50-item questionnaire designed to measure adverse consequences of alcohol abuse in five areas: Interpersonal, Physical, Social, Impulsive, and Intrapersonal. Each scale provides a lifetime and past 3-month measure of adverse consequences, and scales can be combined to assess total adverse consequences. We used a modified version of the DrInC that just included the 45-items that summed the Interpersonal, Physical, Social, and Impulsivity items. This total score (min=0, max=135) was analyzed in this study with high scores indicative of more alcohol-related consequences (a poor outcome for a given study participant). The DrInC was assessed at study weeks 6 and 12. Analyses averaged across these weeks.
Time Frame: Weeks 6 & 12
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Quetiapine Fumerate Plus Medical Management | Sugar Pill Plus Medical Management
Number analyzed (Participants) | 105 | 113
score on a scale | 18.5 (1.87) | 22.5 (1.78)

9. Secondary Outcome: Penn Alcohol Craving Score (PACS_
Description: The Penn Alcohol Craving Scale (PACS) is a five-item, self-report measure that includes questions about the frequency, intensity, and duration of craving, the ability to resist drinking, and asks for an overall rating of craving for alcohol for the previous week (Flannery et al., 1999). The summed total score of the 5 items was used in the analysis (min=0, max=30) with higher scores indicative of higher craving for alcohol (a poor outcome). Based on clinical study results, the PACS has been shown to be a reliable and valid measure of alcohol craving and can predict subjects at risk for subsequent relapse. The PACS was assessed at study weeks 4, 6, 8, 10, and 12. Analyses averaged across these weeks.
Time Frame: Weeks 4, 6, 8, 10, and 12
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Quetiapine Fumerate Plus Medical Management | Sugar Pill Plus Medical Management
Number analyzed (Participants) | 105 | 113
score on a scale | 12.1 (0.63) | 12.8 (0.60)

10. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The MADRS is an observer rating scale that has proven to be an efficient and practical measure of depression (Montgomery and Asberg, 1979). The scale was constructed to be sensitive to changes in treatment effects. Its capacity to differentiate between responders and non-responders to antidepressant treatment has been shown to be comparable to the Hamilton Rating Scale for Depression, another established measure of depressive symptomatology, but the MADRS has greater sensitivity to change during the course of a depressive phase. It has exhibited high inter-rater reliability and appears to be oriented more towards psychic as opposed to somatic aspects of depression. The MADRS is the sum of the 10-item in a checklist where items are rated on a scale of 0 to 6 with anchors at 2-point intervals. Scores range from 0 to 60. Higher scores are indicative of greater depressive symptoms (a poor outcome). The MADRS was assessed at weeks 4, 6, 8, 10, and 12. Analyses averaged across these weeks.
Time Frame: Weeks 3-11
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Quetiapine Fumerate Plus Medical Management | Sugar Pill Plus Medical Management
Number analyzed (Participants) | 105 | 113
score on a scale | 2.8 (0.39) | 4.1 (0.37)

11. Secondary Outcome: Hamilton Anxiety Scale (HAM-A)
Description: The Hamilton Anxiety Scale consists of 14 items, each defined by a series of symptoms. Similar to the HAM-D, each item is rated on a 5-point scale, ranging from 0 (not present) to 4 (severe) (Guy, 1976). A total score is derived from the summed items (min=0, max=56) with higher scores indicative of greater anxiety (a poor outcome). The HAM-A was assessed at study weeks 4, 6, 8, 10, and 12. Analyses averaged across these weeks.
Time Frame: Weeks 4, 6, 8, 10, and 12
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Quetiapine Fumerate Plus Medical Management | Sugar Pill Plus Medical Management
Number analyzed (Participants) | 105 | 113
score on a scale | 2.4 (0.26) | 3.0 (.24)

12. Secondary Outcome: Pittsburgh Sleep Quality Score
Description: The PSQI is a 19-item questionnaire assessing the subject's overall sleep experience in the past 30 days (Buysse et al-1989). The lower the overall score, the better the person sleeps. The tool has an adequate internal reliability, validity and consistency for clinical and community samples of the various populations. Range is (0-21); >6 indicative of "poor" sleep quality. The PSQI was assessed at study weeks 4,8, and 12. Analyses averaged across these weeks.
Time Frame: Weeks 4, 8, 12
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Quetiapine Fumerate Plus Medical Management | Sugar Pill Plus Medical Management
Number analyzed (Participants) | 105 | 113
score | 4.1 (0.27) | 5.1 (0.26)

13. Secondary Outcome: Quality of Life SF - 12 - Mental Aggregate Score
Description: The SF-12 will be used to assess overall health status. The SF-12 is a 12-item questionnaire developed in 1994 as a shorter alternative to the SF-36 to reproduce the physical and mental health summary measures with at least 90% accuracy. We calculated the physical and mental component summary scores which were both converted to T-scores (min=0, max=100) normed to the general population such that a T=50 is the average score in the general population. Higher scores are indicative of better health status.
Time Frame: Week 12
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Quetiapine Fumerate Plus Medical Management | Sugar Pill Plus Medical Management
Number analyzed (Participants) | 105 | 113
score on a scale | 51.5 (1.12) | 50.7 (1.08)

14. Secondary Outcome: Quality of Life SF-12 - Physical Aggregate Score
Description: as for outcome 13
Time Frame: Week 12
Population: mITT
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Quetiapine: Quetiapine fumarate plus medical management
  Quetiapine fumarate: Quetiapine fumarate- taken daily, for 12 weeks
- Placebo: Medical management plus placebo comparator
  Placebo: Placebo
Arm/Group | Quetiapine | Placebo
Number analyzed (Participants) | 105 | 113
score on a scale | 51.0 (0.82) | 50.6 (0.93)

ADVERSE EVENTS:
Description: Systematic assessment at each clinic visit and telephone contact in response to the question "How have you been feeling since the last time we spoke?"
Arm/Group | Quetiapine Fumerate Plus Medical Management | Sugar Pill Plus Medical Management
Serious Adverse Events (participants affected / at risk) | 6/105 | 5/113
Other Adverse Events (participants affected / at risk) | 105/105 | 110/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine Fumerate Plus Medical Management (N=105) | Sugar Pill Plus Medical Management (N=113)
Alcohol Detoxification (Psychiatric disorders) | 3 (4) | 3 (3)
Automobile Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Behavioral Disturbance while intoxicated (Psychiatric disorders) | 0 (0) | 1 (1)
Pre-ventricular contractions (Cardiac disorders) | 0 (0) | 1 (1)
Ruptured Spleen (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine Fumerate Plus Medical Management (N=105) | Sugar Pill Plus Medical Management (N=113)
Dizziness (Nervous system disorders) | 15 (20) | 5 (6)
Dry Mouth (Gastrointestinal disorders) | 34 (36) | 10 (11)
Dyspepsia (Gastrointestinal disorders) | 14 (22) | 2 (2)
Increased Appetite (Metabolism and nutrition disorders) | 12 (12) | 1 (1)
Sedation (Nervous system disorders) | 16 (18) | 3 (3)
Somnelence (Nervous system disorders) | 36 (42) | 10 (10)
Headache (Nervous system disorders) | 36 (60) | 49 (83)
Tremor (Nervous system disorders) | 16 (19) | 14 (18)
Anxiety (Psychiatric disorders) | 20 (26) | 25 (33)
Insomnia (Psychiatric disorders) | 14 (15) | 24 (26)
Depressed Mood (Psychiatric disorders) | 7 (8) | 10 (13)
Abnormal Dreams (Psychiatric disorders) | 10 (10) | 8 (10)
Agitation (Psychiatric disorders) | 10 (11) | 6 (8)
Nausea (Gastrointestinal disorders) | 10 (11) | 20 (25)
Vomiting (Gastrointestinal disorders) | 15 (20) | 14 (15)
Constipation (Gastrointestinal disorders) | 8 (10) | 8 (11)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 11 (12)
Fatigue (General disorders) | 22 (29) | 17 (18)
Feeling Abnormal (General disorders) | 10 (11) | 8 (8)
Irritability (General disorders) | 8 (8) | 7 (9)
Pain (General disorders) | 6 (6) | 9 (9)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 11 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 13 (14)
Oropharynageal Pain (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 6 (7)
Weight Increased (Investigations) | 20 (21) | 12 (13)
Blood Glucose Increased (Investigations) | 3 (3) | 8 (9)
Back Pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 15 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (12) | 5 (6)
Mylagia (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4) | 12 (12)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 (7) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No